CLINICAL TRIAL: NCT03292237
Title: Intensive Nutrition Therapy Compared to Usual Care in Critically Ill Adults: A Randomised Pilot Trial
Brief Title: Intensive Nutrition in Critically Ill Adults
Acronym: INTENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANZIC-RC/ER001
Record Dates: First submitted 2017-09-11; First posted 2017-09-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Critical Illness; Critically Ill
Keywords: Energy; Nutrition; Critical illness; Parenteral nutrition; Intensive care unit; Ward; Randomised Controlled Trial; Intensive Nutrition
MeSH Terms: conditions — Critical Illness; Hyperphagia

STUDY DESIGN:
Intervention Model Description: multicentre, prospective, parallel, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Nutrition Arm (No Intervention): In ICU:
  1. After enrolment, patients allocated to the standard nutrition therapy (control) group will commence or continue nutrition via an enteral tube to a target rate according to unit protocol including the use of promotility agents and the placement of nasojejunal feeding tubes if required.
  2. PN will only be used if the above methods have been attempted, or an absolute contraindication to EN develops.
  3. Unless there is specific indication for a compounded PN solution, the PN used in the standard care group will be the same as used in the intervention arm.
  After ICU:
  1. Nutrition management will be as per usual site management at that hospital.
  2. Nutrition intake amounts will be recorded 3 times per week using provided study documents and assessment tools.
- Intensive Arm (Experimental): Intervention
  In ICU:
  1. Supplemental PN will be commenced within 2 hours of randomisation. The starting dose of PN will be determined by the amount of energy received in the 24 hours prior to randomisation
  2. The need for the intervention will be based on the adequacy of nutrition provision from both PN and EN and assessed daily until ICU discharge
  3. If there is an actual or anticipated interruption of EN for greater than 2 hours the PN must be run at 20 kcal/kg calculated body weight until EN is recommenced. After the interruption, EN should be recommenced as per local protocol.
  After ICU:
  An intensive nutrition intervention will be provided on the ward in the intervention group. This will include daily review from dedicated study dietitians and a clearly protocolized hierarchical management plan which reflects best practice clinical management.
  Interventions: Dietary Supplement: Supplemental parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Supplemental parenteral nutrition — Supplemental parenteral nutrition OLIMEL N12E (Baxter Healthcare Corporation)
  Arms: Intensive Arm

SUMMARY:
Despite the widespread use of nutrition therapy, no large scale randomized controlled trials (RCTs) have demonstrated positive outcomes with delivery of nutrition therapy early in critical illness, with some showing no effect with delayed nutrition or even harm.

There are several possible reasons for the lack of observed benefit from RCTs to date; interventions have been short in duration (usually 3-10 days after intensive care unit (ICU) admission), perhaps applied at the incorrect time in regards to the patients metabolism and recovery, do not consider the patients nutrition risk, and have not addressed what happens to nutrition intake post ICU in critically ill individuals. This may explain why RCTs to date have not observed any positive associations with the delivery of nutrition; our focus to date may have been on the wrong stage of illness. A future study is thus urgently needed, which addresses the deficiencies in current RCTs by optimizing nutrition delivery for the whole hospital stay and collecting meaningful clinical, process and outcome data, which will potentially inform a larger trial of a similar nature.

This initial study aims to determine whether optimization of energy using a pre-tested supplemental parenteral nutrition (PN) strategy in the Intensive Care Unit (ICU) and an intensive nutrition intervention in the post ICU period will deliver more total energy than standard nutrition care during hospital admission in a group of critically ill patients with at least one organ system failure.

DETAILED DESCRIPTION:
Background:

Nutrition is a commonly provided therapy in critical illness, but data about effectiveness is sparse. Best practice guidelines recommend enteral nutrition (EN), a specialised solution delivered into the gastrointestinal tract, as the first line of nutrition therapy. The majority of best practice guidelines also recommend delivery of energy and protein amounts close to predicted requirements in critical illness over the course of Intensive Care Unit (ICU) admission, however the only evidence to support this is from observational data. Although recommended that energy and protein requirements be met, and observational data suggests this is of benefit, there are practical challenges with the provision of EN. International practice surveys report the average energy and protein provided is approximately 59% of the patients predicted requirements, for multifactorial reasons. The addition of parenteral (intravenous) nutrition has been proposed as a method to provide additional energy when EN is insufficient, termed supplemental parenteral nutrition (PN). The ability of this strategy to deliver additional energy and protein to patients during critical illness has been proven in several feasibility/pilot trials, but the benefit on clinical and functional outcomes is unknown.

Despite observational data suggesting benefit when energy and protein delivery is optimised close to requirements, no large scale randomised controlled trials (RCTs) have confirmed improved clinical outcomes in critical illness, with some showing no effect with delayed nutrition or even harm. There are several possible reasons for the lack of observed benefit from RCTs to date; the interventions may have been applied at a time when the patient's metabolism is not in a phase of recovery; interventions have been short in duration and; studies have not addressed what happens to nutrition intake in the post ICU period of hospitalisation in critically ill individuals.

Aims:

To determine whether the use of a pre-tested supplemental PN strategy in the ICU and an intensive nutrition intervention after discharge to the hospital ward is feasible and will deliver more total energy than standard nutrition care over the entire hospital stay, in critically ill patients with at least one organ system failure.

A further aim is to develop a research program that will determine whether optimisation of energy to critically ill patients over the entire period of hospitalisation improves clinically-meaningful outcomes.

Hypothesis:

In critically ill patients with at least one organ failure, the use of a supplemental PN strategy in ICU and an intensive nutrition intervention on the hospital ward will lead to an increase in daily energy delivery of at least 15% over the entire hospital stay when compared to standard care.

Fifteen percent has been estimated as the minimum acceptable clinical difference between the two groups.

Objectives:

The major objectives are:

1. To determine whether the whole hospital nutrition intervention leads to increased amounts of total energy delivered over the period of hospital stay
2. To determine if the whole hospital nutrition intervention is safe in regards to adverse effects
3. To determine if the post-ICU nutrition intervention is practically feasible when applied in multiple hospitals, across multiple wards
4. To measure the clinical outcomes in patients and provide information to assist design of a larger randomised controlled trial

ELIGIBILITY:
Inclusion criteria

Patients in intensive care who meet all of the following will be eligible:

1. Admitted to intensive care between 72 hours and 120 hours
2. Receiving invasive ventilator support
3. At least 18 years of age
4. Have central venous access suitable for PN solution administration
5. Have 1 or more organ system failure (respiratory, cardiovascular or renal) related to their acute illness defined as:

   * PaO2/FiO2 ≤ 300 mmHg
   * Currently on 1 or more continuous inotrope/vasopressor infusion which were started at least 4 hours ago at a minimum dose of:

     1. Noradrenaline ≥ 0.1mcg/kg/min
     2. Adrenaline ≥ 0.1 mcg/kg/min
     3. Any dose of vasopressin
     4. Milrinone > 0.1 mcg/kg/min
   * Renal dysfunction defined as:

     1. Serum creatinine 2.0-2.9 times baseline OR
     2. Urine output 0.5ml/kg/hr for ≥ 12 hours OR
     3. Currently receiving renal replacement therapy
   * Currently has an intracranial pressure monitor or ventricular drain in situ

Exclusion criteria

Patients will be excluded if:

* Both EN and PN cannot be delivered at enrolment (i.e. either an enteral tube or a central venous catheter cannot be placed or clinicians feel that EN or PN cannot be safely administered due to any other reason)
* Currently receiving PN
* Clinician believes a specific parenteral formula is indicated
* Death is imminent in the next 96 hours
* There is a current treatment limitation in place or the patient is unlikely to survive to 6 months due to underlying/chronic illness
* More than 80% of energy requirements have been satisfactorily delivered via the enteral route in the last 24 hours
* Dialysis dependent chronic renal failure
* Suspected or known pregnancy
* Product contraindication
* The treating clinician does not believe the study to be in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Daily energy delivered from nutrition therapy | Day 28
  Daily energy delivered from nutrition therapy

SECONDARY OUTCOMES:
Nutrition intake | Day 28
  Daily protein intake, Energy and protein intake by location (ICU and ward)
Duration hospital stay | Day 28
  Duration of hospital stay in survivors and non-survivors
Ventilator Free Days | Day 28
  Ventilator Free Days (VFDs) at study day 28
Total blood stream infection rate | Day 28
  Total blood stream infection rate

OTHER OUTCOMES:
Duration of ICU stay | Day 28
  Duration of ICU stay in survivors and non survivors
Duration of Mechanical Ventilation | Day 28
  Duration of Mechanical Ventilation to study day 28 in survivors and non-survivors
ICU mobility scale | Day 28
  ICU mobility scale at ICU discharge
Mortality | Day 28
  In hospital and 28 day mortality
Blood stream infections | Day 28
  Number of blood stream infections to day 28, time to any blood stream infection
Weight | Day 28
  Weight at hospital discharge
Frailty | 90 days
  Clinical frailty score
European Quality Of Life 5 Dimensions 5 Level (EQ5D-5L) | 90 days
  Health related quality of life assessment using EQ5D-5L. Each dimension has 5 levels ranging from no problems (1) to extreme problems (5), there is no overall score. It also has a visual analogue scale (VAS) ranging 0-100 with 0 being worst imaginable health state and 100 being best imaginable health state
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 90 days
  WHODAS is a 12 point disability assessment with a raw score range of 0-48. 0 is no disability and 48 being full disability
European Quality Of Life 5 Dimensions 5 Level (EQ5D-5L) | 180 days
  Health related quality of life assessment using EQ5D-5L. Each dimension has 5 levels ranging from no problems (1) to extreme problems (5), there is no overall score. It also has a visual analogue scale (VAS) ranging 0-100 with 0 being worst imaginable health state and 100 being best imaginable health state
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 180 days
  WHODAS is a 12 point disability assessment with a raw score range of 0-48. 0 is no disability and 48 being full disability
Cost per quality adjusted life year | 180 days
  Cost per quality adjusted life year (QALY)
Cost per life year gained | 180 days
  Cost per life year gained (LYG)
Frailty | 180 dyas
  Clinical frailty score

CONTACTS AND LOCATIONS:
Overall Officials: Emma Ridley, PhD, Principal Investigator — ANZIC-RC
Locations (23):
- Australia (21):
  - Blacktown Hospital, Blacktown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Prince Charles Hospital, Brisbane, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Lyell McEwin, Elizabeth Vale, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - Northern Hospital, Epping, Victoria
  - Frankston Hospital - Peninsula Health, Frankston, Victoria
  - Geelong Hospital, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Epworth Richmond, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital CVICU, Auckland
  - Middlemore Hospital, Auckland

IPD SHARING:
Plan to Share IPD: Yes
Data sharing requests will be considered 2 years after publication of the primary trial data on an individual basis by the trial management committee (the data custodians). Data sharing will only be considered for investigator-initiated, independent researchers who provide a written data evaluation proposal that is judged to be methodologically sound. A data sharing agreement will be required to detail conditions under which data is shared and used. Resulting publications should appropriately cite and acknowledge the original data custodians. Requests for data sharing are to be made to anzicrc@monash.edu and the corresponding author, Dr Emma Ridley; emma.ridley@monash.edu

REFERENCES:
- [Derived] Ridley EJ, Bailey M, Chapman MJ, Chapple LS, Deane AM, Gojanovic M, Higgins AM, Hodgson CL, King VL, Marshall AP, Miller EG, McGuinness SP, Parke RL, Paul E, Udy AA; Australian, New Zealand Intensive Care Society Clinical Trials Group. The impact of a tailored nutrition intervention delivered for the duration of hospitalisation on daily energy delivery for patients with critical illness (INTENT): a phase II randomised controlled trial. Crit Care. 2025 Jan 6;29(1):8. doi: 10.1186/s13054-024-05189-3. PMID 39762887
- [Derived] Ridley EJ, Bailey M, Chapman M, Chapple LS, Deane AM, Hodgson C, King VL, Marshall A, Miller EG, McGuinness SP, Parke R, Udy AA; the Australian and New Zealand Intensive Care Society Clinical Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group. Protocol summary and statistical analysis plan for Intensive Nutrition Therapy comparEd to usual care iN criTically ill adults (INTENT): a phase II randomised controlled trial. BMJ Open. 2022 Mar 8;12(3):e050153. doi: 10.1136/bmjopen-2021-050153. PMID 35260448
- [Derived] Ridley EJ. Parenteral nutrition in critical illness: total, supplemental or never? Curr Opin Clin Nutr Metab Care. 2021 Mar 1;24(2):176-182. doi: 10.1097/MCO.0000000000000719. PMID 33315720
- [Derived] Ridley EJ, Parke RL, Davies AR, Bailey M, Hodgson C, Deane AM, McGuinness S, Cooper DJ. What Happens to Nutrition Intake in the Post-Intensive Care Unit Hospitalization Period? An Observational Cohort Study in Critically Ill Adults. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):88-95. doi: 10.1002/jpen.1196. Epub 2018 Jun 20. PMID 29924393